CLINICAL TRIAL: NCT05114798
Title: Effects of Time-restricted Eating Versus Daily Continuous Calorie Restriction on Body Weight and Colorectal Cancer Risk Markers Among Adults With Obesity
Brief Title: Time-restricted Eating Versus Daily Continuous Calorie Restriction on Body Weight and Colorectal Cancer Risk Markers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lisa Tussing-Humphreys, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-1627; 1R01CA257807 (NIH)
Record Dates: First submitted 2021-09-29; First posted 2021-11-10 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Time Restricted Eating; Obesity; Weight Loss; Colorectal Cancer
MeSH Terms: conditions — Intermittent Fasting; Obesity; Weight Loss; Colorectal Neoplasms | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized by the data manager, by way of a stratified random sample in 1:1:1 ratio. The sample frame will be divided into strata based on BMI, sex, and age. Subjects from each stratum, will then be randomized to 1 of 3 groups: 1) TRE, 2) Cal-R, or 3) Control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time Restricted Eating (TRE) (Experimental): During the active weight loss period, the TRE group will be instructed to eat ad libitum from 12:00pm - 8:00pm daily and fast from 8:00pm - 12:00pm. During the 8-h eating window, there will be no restrictions on types or quantities of foods consumed. During the fasting period, participants will be encouraged to drink plenty of water and may consume energy-free beverages, such as black tea or coffee. TRE subjects will meet with the TRE dietitian for 30 minutes at the start of the intervention to review instructions and goals, and then every week throughout the active weight loss period to review intervention adherence. At the beginning of the maintenance phase, total energy needs will be reassessed. Subjects will be instructed to main their body weight by consuming meals in an extended 10-h eating window every day and water fast between 8pm and 10 am, respectively.
  Interventions: Behavioral: Time restricted eating
- Calorie Restriction (Cal-R) (Active Comparator): Cal-R subjects will be instructed to restrict energy intake by 25% of their baseline total energy expenditure (TEE) daily. Subjects will meet with a study dietitian for a 60-min one-on-one session to develop individualized weight loss meal plans to help them adhere to their calorie restriction goal. Meal plans will include portion sizes and food lists that are consistent with their food preferences and prescribed calorie levels for weight loss. Food scales will be provided to help with food portioning. Cal-R subjects will meet with the dietitian every week throughout the weight loss period to review intervention adherence and modify the meal plans as needed. Subjects will be asked to maintain their baseline level of physical activity. At the beginning of the weight maintenance phase, total energy needs will be reassessed.
  Interventions: Behavioral: Calorie Restriction
- Control (No Intervention): Controls will be instructed to maintain their weight throughout the 12 m trial and to not change eating or physical activity habits. Controls will not receive dietary counseling. Controls will visit the research center every 3 months for outcome measurements.

INTERVENTIONS:
Behavioral: Time restricted eating — daily ad libitum food intake, 8-h 12pm - 8pm, 6 m active weight loss phase; 10-h 10am-8pm, 6 m maintenance phase
  Arms: Time Restricted Eating (TRE)
Behavioral: Calorie Restriction — daily 25% calorie restriction, 6 m active weight loss phase; 100% energy needs, 6 m maintenance phase
  Arms: Calorie Restriction (Cal-R)

SUMMARY:
Approximately 42% of American adults are obese, and this condition is strongly related to the development of colorectal cancer. Innovative lifestyle strategies to treat obesity and reduce colorectal cancer risk are critically needed. This research will demonstrate that time-restricted eating, a type of intermittent fasting, is an effective therapy to help obese individuals reduce and control their body weight and prevent the development of colorectal cancer.

DETAILED DESCRIPTION:
Approximately 42% of the U.S. adult population is obese and data suggests that persons with obesity are at a 30% greater risk of developing colorectal cancer (CRC). Therefore, efficacious approaches to preventing and treating obesity will have significant effects on CRC incidence in the U.S. Although calorie restriction through lifestyle intervention is the most common approach to treat obesity, clinically meaningful weight loss is difficult to achieve via this method due to low adherence with calorie monitoring, indicating a need for innovation. Time-restricted eating, a type of intermittent fasting, has been shown in animals to impart cancer protective effects including lower body weight, decreased systemic inflammation, and improved glucose metabolism. Time-restricted eating is where individuals are asked to consume all their food for the day within a specified time frame, and water fast for the remaining hours of the day. We recently performed two short-term (≤12-weeks) pilot studies of time-restricted eating to evaluate its safety and preliminary efficacy on body weight and chronic disease risk markers in adults with obesity. Our results show the intervention is a safe and acceptable approach to weight loss among obese adults. Moreover, time-restricted eating produced approximately 3% weight loss from baseline and reductions in systolic blood pressure, oxidative stress and insulin resistance. Although these pilot findings show promise for time-restricted eating as an effective tool for CRC risk reduction among obese individuals, these data still require confirmation by a well powered longer-term clinical trial. The present proposal aims to implement a 12-month (6-month intervention, 6-month maintenance) controlled, parallel arm trial among 255 obese adults (45-70 years old) who have had a colonoscopy. Subjects will be randomized to 1 of 3 groups: 1) 8-hour time-restricted eating (daily ad libitum food intake from 12pm - 8pm), 2) Calorie restriction (daily 25% calorie restriction), or 3) Control (daily ad libitum food intake, no meal timing restrictions) to compare the effects on: (1) Body weight, body composition, and intervention adherence; (2) Circulating metabolic, inflammation, and oxidative stress-related biomarkers; (3) Colonic mucosal gene expression profiles and mucosal inflammation, DNA damage and cellular growth; and (4) maintenance of benefits on body weight/composition and CRC markers.

ELIGIBILITY:
Inclusion Criteria:

1. 45-70 years old,
2. BMI 30-49.99 kg/m2
3. Are up to date with CRC screening.

Exclusion Criteria:

1. Have a history of renal disease, autoimmune disorders, immunodeficiency, malabsorptive disorder, significant gastrointestinal and hepatic disease, surgical change in gastrointestinal anatomy, severe ischemic heart disease, severe pulmonary disease, severe mental health disorder, eating disorder, or bariatric surgery;
2. Abuse alcohol (> 50 grams/day), illicit drugs (other than self-reported marijuana use), or use combustible tobacco;
3. Have controlled type 2 diabetes or undiagnosed uncontrolled diabetes based on hemoglobin A1c (HbA1c) > 9.0%;
4. Have a history of cancer treatment within the past 12 months, CRC, genetic predisposition to CRC (e.g., Lynch syndrome);
5. Have a baseline body weight > 450 lbs (weight limitation of the DXA);
6. Are on a weight loss diet or actively involved in a formal weight loss program (e.g., Weight Watchers);
7. Are not weight stable for 3 months prior to the study (weight gain or loss > 4 kg);
8. Are unable to keep a food diary for 7 consecutive days during screening;
9. Are night shift workers;
10. Are pregnant or trying to get pregnant;
11. Are taking drugs that influence study outcomes (weight loss medications);
12. Are non-English speaking
13. Are taking anticoagulant medications or medications with endoscopic risk
14. Are taking antivirals or immunosuppressant medications
15. Don't have regular access to an email address and computer/smartphone/tablet
16. Are currently following a diet that requires fasting on a weekly basis
17. Currently eat for less than 10 hours of the day (determined by asking participants what time they start and stop eating on a usual day)

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Weight change (% kg) | Baseline to month 6
  Body weight in kg

SECONDARY OUTCOMES:
Total and regional body fat composition and distribution | Baseline, 6 month and 12 month
  Total and regional body fat composition and distribution will be measured via whole body DEXA scan
Intervention adherence | Monthly, through month 6
  Measured through electronic diet records and 24 hour dietary recalls
Fasting plasma glucose | Baseline, month 3, month 6, month 9, month 12
  From fasting venous blood measured by a commercial lab
Plasma cytokines TNF-α, IL-6, IL1-β, and IL-10, % | Baseline, month 3, month 6, month 9, month 12
  Multiplex ELISA
Plasma 8-isoprostane | Baseline, month 3, month 6, month 9, month 12
  ELISA
Colonic mucosa gene expression profiling | Baseline, month 6, month 12
  Commercially available targeted transcriptomics platform
Ki-67, proliferation | Baseline, month 6, month 12
  Healthy colonic mucosa, immunohistochemistry
c-caspase-3, Bax, apoptosis | Baseline, month 6, month 12
  Healthy colonic mucosa, immunohistochemistry,
CD3, CD163, pIKKa/b, tissue markers of inflammation | Baseline, month 6, month 12
  Healthy colonic mucosa, immunohistochemistry
Weight maintenance (% kg) | Month 6 to month 12
  Maintenance of weight loss
Fasting plasma insulin | Baseline, month 3, month 6, month 9, month 12
  From fasting venous blood measured at a commercial lab
HOMA-IR | Baseline, month 3, month 6, month 9, month 12
  calculated from fasting glucose and insulin using a standard formula
Gut Microbiome | Baseline, month 3 and month 6
  Shotgun metagenomics
Fecal Metabolites | Baseline, month 3 and month 6
  Untargeted Metabolomics
Saliva microbiota | Baseline, month 3, month 6
  Untargeted Metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Tussing-Humphreys, PhD, MS, RD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No